CLINICAL TRIAL: NCT03373630
Title: Prospective Analysis of Incidence and Risk Factors of Infection of Midline Catheter
Acronym: TIM-GHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Collaborators: TIMC-IMAG (Other); Vygon GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/11-DFO-GHMG
Record Dates: First submitted 2017-11-23; First posted 2017-12-14 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Intravascular Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midline catheter (Experimental)
  Interventions: Device: Midline catheter

INTERVENTIONS:
Device: Midline catheter — The catheter will be inserted according to usual practices, after the enrollment of the patient in the study. The follow-up will last until the removal of the catheter, which will also be done according to usual practices. Following the removal, bacteriologic analyses will be performed in order to diagnose any prospective infection.

SUMMARY:
The Midline catheter is a peripherally-inserted catheter, with the distal tip being placed at or below the level of the axilla. It is a relevant alternative to other catheters in case of limited venous access and long-run perfusions. Moreover, another significant advantage may be the reduction of the risk of infection.

However, the Midline catheter is poorly described in scientific literature, essentially through retrospective and meta analyses including multiple types of catheters (Piccline, CVC, PAC). Therefore, the TIM-GHM study aims to prospectively assess the rate of infections in case of the Midline catheter.

The results of this study could bring a collective benefit in terms of knowledge and reliability of these intravascular devices.

Depending on these results, a randomized, controlled study will be considered, in order to compare the Midline catheter to its main alternative : the Piccline.

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal to 18 years old
* Intravascular treatment planned for more than 6 days

Exclusion Criteria:

* Medical history of mastectomy with bilateral lymphadenectomy
* Peripheral neuropathy
* Upper-Extremity Deep Vein Thrombosis
* Arteriovenous fistula
* Poor condition of the skin of the upper limbs
* Patient in palliative care
* Patient in emergency care
* Patient under guardianship/curatorship
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of infection of midline catheter | Catheter removal, performed up to 28 days after enrollment
  The method used for bacteriologic analyses will be the Brun Buisson Technique. The diagnosis of infection of the catheter will be based on the clinical signs, the catheter bacteriology, the blood culture collected on the patient and the blood culture collected on the catheter.

SECONDARY OUTCOMES:
Identification of the germs responsible for infections of midline catheter | Catheter removal, performed up to 28 days after enrollment
  For each infected catheter, the species name of the germ responsible for the infection will be collected.
Identification of intravenous treatments - Corticosteroid | Everyday from baseline, up to 28 days
  Determination of whether corticosteroid are intravenously administered during the day (YES/NO).
Identification of intravenous treatments - Antibiotics | Everyday from baseline, up to 28 days
  Determination of whether antibiotics are intravenously administered during the day (YES/NO).
Identification of intravenous treatments - Chemotherapy | Everyday from baseline, up to 28 days
  Determination of whether chemotherapy was intravenously administered during the day (YES/NO).
Identification of intravenous treatments - Nutrient solution | Everyday from baseline, up to 28 days
  Determination of whether nutrient solution was intravenously administered during the day (YES/NO).
Duration of insertion procedure | Baseline
Lifetime of catheter | Catheter removal, performed up to 28 days after enrollment
  Time from catheter insertion to catheter removal, measured in days.
Body Mass Index | Baseline
White blood cells count | Everyday from baseline, up to 28 days
Incidence of thrombosis | Catheter removal, performed up to 28 days after enrollment
  If the catheter is no more permeable, a doppler echocardiography will be done to confirm the diagnosis of thrombosis.
Patient comfort | Every three days from baseline, up to 28 days
  Numeric rating scale will be collected for each of these 3 dimensions : comfort when eating, comfort when moving, comfort for personal hygiene The scale will range from 0 to 10. 0 will mean "very uncomfortable" and 10 will mean "very comfortable".

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Mutualiste de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goetz AM, Miller J, Wagener MM, Muder RR. Complications related to intravenous midline catheter usage. A 2-year study. J Intraven Nurs. 1998 Mar-Apr;21(2):76-80. PMID 9601314
- [Background] Chopra V, Ratz D, Kuhn L, Lopus T, Chenoweth C, Krein S. PICC-associated bloodstream infections: prevalence, patterns, and predictors. Am J Med. 2014 Apr;127(4):319-28. doi: 10.1016/j.amjmed.2014.01.001. Epub 2014 Jan 17. PMID 24440542
- [Background] Timsit JF, Dubois Y, Minet C, Bonadona A, Lugosi M, Ara-Somohano C, Hamidfar-Roy R, Schwebel C. New materials and devices for preventing catheter-related infections. Ann Intensive Care. 2011 Aug 18;1:34. doi: 10.1186/2110-5820-1-34. PMID 21906266
- [Background] Ugas MA, Cho H, Trilling GM, Tahir Z, Raja HF, Ramadan S, Jerjes W, Giannoudis PV. Central and peripheral venous lines-associated blood stream infections in the critically ill surgical patients. Ann Surg Innov Res. 2012 Sep 4;6(1):8. doi: 10.1186/1750-1164-6-8. PMID 22947496
- [Background] Ziegler MJ, Pellegrini DC, Safdar N. Attributable mortality of central line associated bloodstream infection: systematic review and meta-analysis. Infection. 2015 Feb;43(1):29-36. doi: 10.1007/s15010-014-0689-y. Epub 2014 Oct 21. PMID 25331552
- [Background] Zochios V, Umar I, Simpson N, Jones N. Peripherally inserted central catheter (PICC)-related thrombosis in critically ill patients. J Vasc Access. 2014 Sep-Oct;15(5):329-37. doi: 10.5301/jva.5000239. Epub 2014 Apr 25. PMID 24811591
- [Background] Mermel LA, Parenteau S, Tow SM. The risk of midline catheterization in hospitalized patients. A prospective study. Ann Intern Med. 1995 Dec 1;123(11):841-4. doi: 10.7326/0003-4819-123-11-199512010-00005. PMID 7486466
- [Background] Pongruangporn M, Ajenjo MC, Russo AJ, McMullen KM, Robinson C, Williams RC, Warren DK. Patient- and device-specific risk factors for peripherally inserted central venous catheter-related bloodstream infections. Infect Control Hosp Epidemiol. 2013 Feb;34(2):184-9. doi: 10.1086/669083. Epub 2012 Dec 14. PMID 23295565